CLINICAL TRIAL: NCT02048462
Title: The Effect of Strenuous Exercise on Coagulation: Hemostatic Behaviour Before and After Amstel Gold Race
Brief Title: The Effect of Strenuous Exercise on Coagulation.
Status: Completed | Type: Observational
Sponsor: Synapse bv (Industry)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL47367.068.13
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: The Effect of Strenuous Exercise on Haemostasis.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cyclists

SUMMARY:
Many studies have shown that vigorous exercise increases the risk of developing vascular thrombotic events and can result in sudden death during or immediately after exercise. The outcome of these studies is biased by several confounding variables: subjects, type of exercise, duration, intensity and especially the method used for the evaluation of the hemostatic capacity. The goal of our study is to investigate the effect of strenuous exercise with the Calibrated Automated Thrombogram (CAT) assay, which is an established tool in detecting hyper- and hypocoagulabilty conditions. We modified the CAT assay to make it also feasible to measure TG in whole blood (WB-CAT), not only to go one step closer to physiology since all the blood cells are present, but also to avoid the centrifugation step. With our study we would like to see whether the other blood cells also play a role in the increase in TG. The objective is to investigate the effect of strenuous exercise (participation to the Amstel Gold Race) on coagulation and haemostatic parameters. We hypothesize that strenuous exercise induces a prothrombotic phenotype and that especially the tests involving blood cells will be altered into a prothrombotic phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects not taking any medication interfering with coagulation that are willing to donate 18 ml of blood via venipuncture and a capillary blood drop via fingerpuncture before and after the Amstel Gold Race.
* Between 18 and 50 years of age. We take 50 year as a maximal age to prevent any co-morbidity that could have an influence on coagulation (like diabetes, atherosclerosis, peripheral arterial disease, …).

Exclusion Criteria:

* Subjects taking any medication interfering with coagulation.
* Subjects having a cardiovascular disease or any other serious medical problem.
* Subjects below 18 years or above 50 years of age.
* Subjects that smoke.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants of the Amstel Gold Race for non-professionals will be asked to join our study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The effect of strenuous exercise on thrombin generation and other coagulation tests. | Before and after the Amstel Gold Race (around 6 hours)
  Thrombin generation will be done in whole blood and plasma. The parameters we will study at are: the peak height, ETP, lagtime, time-to-peak and velocity index.
  Routine coagulation tests (APTT, PT, INR, platelet count, haematocrit, fibrinolysis assay, FACS, ROTEM, ABO-determination, dRVVT-X, D-dimers) Measurements of coagulations factor levels (II, V, VII, VIII, IX, X, XI, XII, fibrinogen, protein S and C, ADAMTS-13)

CONTACTS AND LOCATIONS:
Locations (1):
- Synapse bv, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Huskens D, Roest M, Remijn JA, Konings J, Kremers RM, Bloemen S, Schurgers E, Selmeczi A, Kelchtermans H, van Meel R, Meex SJ, Kleinegris MC, de Groot PG, Urbanus RT, Ninivaggi M, de Laat B. Strenuous exercise induces a hyperreactive rebalanced haemostatic state that is more pronounced in men. Thromb Haemost. 2016 Jun 2;115(6):1109-19. doi: 10.1160/TH15-10-0821. Epub 2016 Feb 11. PMID 26864794